CLINICAL TRIAL: NCT06435052
Title: Efficacy of Eye Movement Desensitization & Reprocessing vs Cognitive Behavioral Therapy in Post-Traumatic Stress and Comorbid Disorders in Pakistan: A Full-fledged Randomized Controlled Trial
Brief Title: Efficacy of Eye Movement Desensitization & Reprocessing vs Cognitive Behavioral Therapy in Post-Traumatic Stress and Comorbid Disorders in Pakistan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khushal Khan Khattak Univeristy, Karak, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Anwar Khan, Dr. Anwar Khan, Assistant Professor of Organizational Psychology, Khushal Khan Khattak Univeristy, Karak, Pakistan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 111
Record Dates: First submitted 2023-02-01; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Post Traumatic Stress Disorder; Depression, Anxiety
Keywords: Post Traumatic Stress Disorder; EMDR; CBT; Pakistan
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization & Reprocessing Therapy (Experimental): Eye Movement Desensitization and Reprocessing (EMDR) therapy will be administered face-to-face by a psychotherapist in a total of 12 sessions, with one session per week. The efficacy of EMDR therapy will be compared with Cognitive Behavioral Therapy (CBT) in the treatment of Post-Traumatic Stress Disorder (PTSD) in Pakistan.
  Interventions: Behavioral: Eye Movement Desensitization & Reprocessing Therapy
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy (CBT) will be delivered face-to-face by a psychotherapist in a total of 14 sessions, with one session per week. The efficacy of CBT will be compared with Eye Movement Desensitization and Reprocessing therapy in the treatment of Post-Traumatic Stress Disorder in Pakistan.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Eye Movement Desensitization & Reprocessing Therapy — Eye Movement Desensitization and Reprocessing (EMDR) therapy will be administered face-to-face by a psychotherapist in a total of 12 sessions, with one session per week. The efficacy of EMDR therapy will be compared with Cognitive Behavioral Therapy in the treatment of Post-Traumatic Stress Disorder in Pakistan.
  Arms: Eye Movement Desensitization & Reprocessing Therapy
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy will be comparatively checked with Eye Movement Desensitization & Reprocessing Therapy for its efficacy. It will be administered by psychotherapist in 14 sessions (each session per week)
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This Randomized Controlled Trial will check the efficacy of Eye Movement Desensitization & Reprocessing vs Cognitive Behavioral Therapy in Post-Traumatic Stress and Comorbid Disorders in Pakistan

DETAILED DESCRIPTION:
This Randomized Controlled Trial will check the efficacy of Eye Movement Desensitization & Reprocessing vs Cognitive Behavioral Therapy in Post-Traumatic Stress and Comorbid Disorders in Pakistan.

It will be a single blind multi-center RCT with two arms (EMDR and CBT). This study will broadly work on following aims:

1. Initially the comparative efficacy of EMDR and CBT (i.e., standard face-to-face protcols) will be determined on large scale in Pakistan by:

   1. Examining whether EMDR is non-inferior to CBT in the treatment of PTSD and its two comorbidities in Pakistan.
   2. Studying changes in the symptoms (i.e., reduction in the PTSD and comorbid symptoms with the passage of time) after administering EMDR and CBT. The level of change in the symptoms will ultimately help in determining the extent of effectiveness of both therapies.
   3. Examine the reciprocal relationship between PTSD and comorbid symptoms for knowing whether any reduction in the PTSD symptoms can help in reducing the comorbid symptoms after administering EMDR and CBT.
2. At the mean time work on the design and development of virtual EMDR and CBT therapies (i.e., Web-based and Mobile Applications) will also be started. The initial prototypes will be tested for its comparative efficacy. Later once the final versions will be developed then it will be also tested for its comparative efficacy on large scale in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

reverse of the exclusion critera

Exclusion Criteria:

The following patients will be excluded:

1. Patients below the age of 15 years and above 60 years, since this study is neither on children nor on old aged patients;
2. Patients who can't move their hands and eyes/or can't perform basic movements;
3. Patients who are unconscious for longer periods and unable to recover consciousness;
4. Patients not meeting the basic screening criteria of PTSD/ PTSD is not the main problem;
5. Patients with severe intellectual impairments, since such patients are difficult to communicate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder | 2 years
  Post-traumatic stress disorder (PTSD) will be assessed using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). The CAPS-5 scores will be utilized to determine the severity of PTSD symptoms. Typically, a CAPS-5 score of 40 or above will serve as the cutoff point for diagnosing PTSD.

SECONDARY OUTCOMES:
Depressive and Anxiety Symptoms | 2 years
  Depressive and anxiety symptoms will be measured using the Hamilton Depression Rating Scale and the State-Trait Anxiety Inventory, respectively. A Hamilton Depression Rating Scale score of 20 or above, and a State-Trait Anxiety Inventory score of 40 or above, will serve as the cutoff points.

CONTACTS AND LOCATIONS:
Locations (1):
- Anwar Khan, Karak, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
can be shared on request